CLINICAL TRIAL: NCT03904004
Title: Impact of Peroral Endoscopic Myotomy and Other Treatments for Oesophageal Motility Disorders on Bolus Transport and Gastro-oesophageal Reflux. The pFlow Study
Brief Title: Pressure and Flow Study Before and After Treatments for EMD. The pFlow Study
Acronym: pFlow
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: EST-ALB-pFlow
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Esophageal Motility Disorders; Gastro-esophageal Reflux
Keywords: esophageal motility disorders; laparoscopic Heller myotomy; peroral endoscopic myotomy; neumatic cilatation; botulinic toxin injection; gastro esophageal reflux
MeSH Terms: conditions — Esophageal Motility Disorders; Gastroesophageal Reflux | interventions — Botulinum Toxins; Botulinum Toxins, Type A; Heller Myotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Esophageal motility disorders: Individuals with sympmtoms related to esophageal motility disorders who receive a endoscopic or surgical treatment
  Interventions: Procedure: Peroral endoscopic myotomy; Procedure: Neumatic dilatation; Procedure: Botulinum toxin injection; Procedure: Laparoscopic Heller Myotomy

INTERVENTIONS:
Procedure: Peroral endoscopic myotomy — Endoscopic myotomy after performing a tunnel to reach the muscular layer through a mucosal incision
  Other Names: POEM
Procedure: Neumatic dilatation — Inflation of a ballon of specific diameter in the gastro-oesophageal junction
Procedure: Botulinum toxin injection — Injection of botulinic toxin to inhibit the contraction of the gastro-oesophageal junction muscular layer
  Other Names: Botox
Procedure: Laparoscopic Heller Myotomy — Five or six small incisions are made in the abdominal wall and laparoscopic instruments are inserted. The myotomy is a lengthwise cut along the oesophagus, starting above the lower oesophageal sphincter (LOS) and extending down onto the stomach a little way. The oesophagus is made of several layers, and the myotomy only cuts through the outside muscle layers which are squeezing it shut, leaving the inner mucosal layer intact.

SUMMARY:
Pressure and flow (PF) analysis allow a detailed report on the bolus passing for each segment of the esophagus. This approach has evidence in oropharyngeal dysphagia, post reflux surgery dysphagia, gastroesophageal reflux in infants and dysphagia in patients with normal manometry. However, it has not been used for defined esophageal motility disorders and their response to surgical or endoscopic treatments. Better knowledge about pre and postoperative bolus flow can yield important concepts that can modify the selection of optimal treatments.

DETAILED DESCRIPTION:
Methods This is an international multicenter prospective observational study in a cohort of individuals affected by an oesophageal motor disorder (OMD).

Participating centers OMD are treated in most tertiary hospitals surgically (Laparoscopic Heller Myotomy (LHM)) or endoscopically (botulinic toxin injection, pneumatic dilatation or peroral endoscopic myotomy (POEM)). The main requirement is to perform high-resolution manometry with impedance before and after the procedure.

Subjects Inclusion criteria are to present with gastrointestinal (GI) symptoms that are secondary to OMD such as dysphagia, regurgitation and/or non-cardiac chest pain. OMD under study are achalasia type I, II and III; oesophagogastric junction (OGJ) outflow obstruction; distal oesophageal spasm, hypercontractile oesophagus or disorders not fulfilling Chicago Criteria version 3. Treatments included are outlined in the previous paragraph.

Exclusion criteria are the inability to fill in symptom questionnaires, intolerance of pre or postprocedure test, incomplete therapeutic procedures or artifacts in manometry/impedance tracings.

Data sharing High-resolution manometry (HRM)-impedance studies will be shared and PF analysis will be performed through Swallow Gateway®. See Appendix 1 for further detail. An acrobat sheet will be eased to fill-in symptomatic and test data pre and post-procedure. It will also be shared through Swallowgateway®.

Variables

1. Demographics: age, sex, anesthetic risk assessment (ASA), height and weight, proton pump inhibitors (PPI) intake.
2. Previous treatments:

   1. Type of treatment.
   2. Number of previous treatments.
   3. Years before current treatment.
3. Symptoms: time from symptoms onset, dysphagia scores (Eckardt, Mellow-Pinkas), gastro-esophageal reflux score questionnaire (GERD-Q), heartburn and regurgitation visual analogic score (VAS), quality of life score short form 12 (SF-12).
4. Pre and post-operative test:

   1. Endoscopy: sigmoid oesophageal dilatation, solid/liquid oesophageal remanent, difficulty to progress through OGJ, oesophagitis (Los Angeles score).
   2. Barium swallow: oesophageal diameter [grade I (< 3.5 cm), grade II (3.5-6 cm) and grade III (> 6 cm)]14, barium column height at 1 and 5 min post-swallowing.
   3. High-resolution manometry: equipment specification (probe, system), morphologic classification of the OGJ, end-expiratory basal pressure, 4 second integrated relaxation pressure (4s-IRP), mean distal contractile integrity (DCI), percentage of failed swallows (DCI<100 mmHg-cm-s), distal latency (DL), percentage of swallows with distal oesophagus pressurization > 30 mmHg, percentage of swallows with pan oesophageal pressurization, type of peristalsis after rapid swallow test, pan oesophageal pressurization after multiple swallow test. Chicago v3 diagnosis of motility pattern.
5. Procedure variables:

   a. Botulinic toxine: i. International units (IU) delivered. ii. Number of toxine injection sessions. iii. Region of oesophagus where the toxin is injected. iv. Complications description, severity and management*. b. Pneumatic dilatation: i. Size of the balloon. ii. Number of dilatations. iii. Complications description, severity and management *. iv. In-hospital stay length**. c. POEM: i. Number of POEM performed by the endoscopist. ii. Anterior or posterior approach. iii. Oesophageal tunnel length. iv. Gastric tunnel length. v. Oesophageal myotomy length. vi. Gastric myotomy length. vii. Full-thickness or partial myotomy. viii. Duration of the procedure. ix. Complications description, severity and management *. x. In-hospital stay length**. d. Laparoscopic Heller Myotomy: i. Number of LHM performed by the surgeon. ii. Oesophageal myotomy length. iii. Gastric myotomy length. iv. Duration of the procedure. v. Complications description, severity and management*. vi. In-hospital stay length**.
6. Pre and post-operative pressure-flow analysis in HRM-impedance:

   - HRM-impedance protocol: patient preparation and HRIM catheter insertion are recommended as described previously (see references) in a recumbent and an inclination of 0 to 30 degrees of head elevation. After positioning of the probe sensors and a 5-min rest period, swallow-induced peristalsis will be tested at 30s intervals. Ten 5-mL liquid swallows (0.9% saline) will be delivered. Peristalsis recovery (weak or normal peristalsis in > 1 swallow with normal DL).

   a. Three measures of intra-bolus distension pressures (DP) during bolus transport were determined at nadir impedance7. These pressures were i. DP bolus accommodation (DPA), intra-bolus distension pressure recorded between the upper oesophageal sphincter (UOS) and the transition zone (TZ); ii. DP compartmentalized transport (DPCT), intra-bolus distension pressure recorded between the TZ and the contractile deceleration point, (CDP); and iii. DP during oesophageal emptying (DPE), intra-bolus distension pressure recorded between the CDP and crural diaphragm (CD).

   b. Bolus clearance from the oesophagus was determined by the impedance ratio (IR = oesophageal nadir impedance divided by impedance recorded during contractile peak pressure). Higher IR indicates less effective oesophageal clearance16.

   c. Two measures of bolus flow latencies, determined at the CDP level, were i. swallow initiation to maximal bolus distension latency (SDL) and ii. maximal bolus distension to contraction latency (DCL). d. Pressures generated during bolus clearance (or clearance pressures) were measured within the distal oesophagus. The closure pressure (CP) was the pressure at luminal closure and the rate of ramp pressure (RP) was the mean gradient of pressure during closure. Timing of luminal closure was taken as when impedance had recovered 50 %, a validated criterion in widespread use17.

   e. A pressure-flow index (PFI) composite score was derived using the following formula: PFI = (DPE*RP)/DCL i.e. the distal IBP during the phase of oeosphageal emptying multiplied by the rate of ramp pressure rise, divided by the time interval from bolus distension to contraction latency.

   f. Bolus presence time (BPT) was estimated based on the method of Lin within the 2 cm segment above the CD landmark.

   g. Trans-OGJ bolus flow time (BFT) was calculated also according to the method of Lin, recording the time deemed favourable for bolus flow across the OGJ.
7. 24h pH/impedance testing.

   * Following American Society for gastrointestinal endoscopy (ASGE) lexicon. **Days after finishing the procedure.

Analysis Main outcome

1. Compare the modification of PF variables between the type of treatment groups for the same OMD.

Secondary outcomes

1. Comparison of pre-procedure PF variables within patients diagnosed with the same manometric subtype.
2. Correlation of PF variables before and after treatment with the respective symptoms.
3. Comparison of post-procedure PF variables between patients with clinical success and clinical failure.
4. Correlation of post-procedure PF variables with barium column.
5. Comparison of post-procedure PF variables between patients with and without post-procedure GOR.
6. Correlation of post-procedure PF variables with grade of Los Angeles oesophagitis classification, % of distal oesophageal acid exposure time and deMeester score.

Visits protocol Visit 1 - at pre-procedure HRM impedance

* Delivery of informed consent.
* Demographic and symptomatic data interrogation.
* Gather endoscopy and barium swallow data.
* HRM impedance testing.
* Procedure choice and explanation. Visit 2 - at hospital discharge
* Procedure-related variables.
* Complications.
* In-hospital stay length. Visit 3 - 3 to 6 months post-procedure
* Symptom-related data.
* Endoscopy and barium swallow data.
* HRM impedance testing.
* 24h pH/impedance testing.
* Data sharing through Swallow Gateway®. Visit 4 - 1 year post-procedure
* Symptomatic data interrogation

ELIGIBILITY:
Inclusion Criteria:

* to present with GI symptoms that are secondary to EMD such as dysphagia, regurgitation and/or non-cardiac chest pain.
* the EMD patients to be recruited under this study are achalasia type I, II and III; OGJ outflow obstruction; distal oesophageal spasm, hypercontractile oesophagus or disorders not fulfilling Chicago Criteria v3.
* Receive a treatment such as POEM, neumatic dilatation, LHM, botox injection.

Exclusion Criteria:

* Exclusion criteria are the inability to fill in symptom questionnaires, intolerance of pre or post procedure test, incomplete therapeutic procedures or technical failure of baseline manometry investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age and sex diagnosed with an EMD that generate symptoms
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Bolus Pressure and Flow (PF) modification | 6 months
  Compare oesophageal biomechanics (based on PF analysis) before and after the different surgical or endoscopic treatments for oesophageal motility disorders (OMD). This analysis describes through numeric variables the passing of the bolus from the mouth to the stomach regarding resistance of flow, clearance and velocity for every part of the oesophagus

SECONDARY OUTCOMES:
PF analysis within similar OMD | 6 months
  Compare PF variables (as described in Outcome 1) within the same OMD at the moment previously to the treatment.
Symptom correlation | 12 months
  Correlate PF variables with pre and post-treatment symptoms of dysphagia, chest pain, regurgitation and heartburn symptom scoring.
Clinical success correlation | 12 months
  Identify PF variables that may be predictors with clinical success and failure as described in the symptom scoring tests.
Correlation with barium column | 6 months
  Identify PF variables that are predictors of timed barium column as a surrogate of prognosis
Correlation with reflux | 6 months
  Identify PF variables that are predictors of post-procedure gastro-oesophageal reflux (GOR) diagnosis after endoscopy - regarding oesophagitis- and 24h pH test -regarding percentage of distal oesophagus acid exposure and deMeester score.

CONTACTS AND LOCATIONS:
Overall Officials: Fermin Estremera-Arevalo, MD, PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Estremera-Arevalo F, Albeniz E, Rullan M, Areste I, Iglesias R, Vila JJ. Efficacy of peroral endoscopic myotomy compared with other invasive treatment options for the different esophageal motor disorders. Rev Esp Enferm Dig. 2017 Aug;109(8):578-586. doi: 10.17235/reed.2017.4773/2016. PMID 28617027
- [Background] Khashab MA, Familiari P, Draganov PV, Aridi HD, Cho JY, Ujiki M, Rio Tinto R, Louis H, Desai PN, Velanovich V, Albeniz E, Haji A, Marks J, Costamagna G, Deviere J, Perbtani Y, Hedberg M, Estremera F, Martin Del Campo LA, Yang D, Bukhari M, Brewer O, Sanaei O, Fayad L, Agarwal A, Kumbhari V, Chen YI. Peroral endoscopic myotomy is effective and safe in non-achalasia esophageal motility disorders: an international multicenter study. Endosc Int Open. 2018 Aug;6(8):E1031-E1036. doi: 10.1055/a-0625-6288. Epub 2018 Aug 10. PMID 30105290
- [Background] Schlottmann F, Luckett DJ, Fine J, Shaheen NJ, Patti MG. Laparoscopic Heller Myotomy Versus Peroral Endoscopic Myotomy (POEM) for Achalasia: A Systematic Review and Meta-analysis. Ann Surg. 2018 Mar;267(3):451-460. doi: 10.1097/SLA.0000000000002311. PMID 28549006
- [Background] Kane ED, Budhraja V, Desilets DJ, Romanelli JR. Myotomy length informed by high-resolution esophageal manometry (HREM) results in improved per-oral endoscopic myotomy (POEM) outcomes for type III achalasia. Surg Endosc. 2019 Mar;33(3):886-894. doi: 10.1007/s00464-018-6356-0. Epub 2018 Jul 27. PMID 30054739
- [Background] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJ, Pandolfino JE; International High Resolution Manometry Working Group. The Chicago Classification of esophageal motility disorders, v3.0. Neurogastroenterol Motil. 2015 Feb;27(2):160-74. doi: 10.1111/nmo.12477. Epub 2014 Dec 3. PMID 25469569
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Bredenoord AJ, Hebbard GS. Technical aspects of clinical high-resolution manometry studies. Neurogastroenterol Motil. 2012 Mar;24 Suppl 1:5-10. doi: 10.1111/j.1365-2982.2011.01830.x. PMID 22248102
- [Background] Imam H, Shay S, Ali A, Baker M. Bolus transit patterns in healthy subjects: a study using simultaneous impedance monitoring, videoesophagram, and esophageal manometry. Am J Physiol Gastrointest Liver Physiol. 2005 May;288(5):G1000-6. doi: 10.1152/ajpgi.00372.2004. PMID 15826930
- [Result] Nguyen NQ, Holloway RH, Smout AJ, Omari TI. Automated impedance-manometry analysis detects esophageal motor dysfunction in patients who have non-obstructive dysphagia with normal manometry. Neurogastroenterol Motil. 2013 Mar;25(3):238-45, e164. doi: 10.1111/nmo.12040. Epub 2012 Oct 31. PMID 23113942
- [Result] Singendonk MM, Kritas S, Cock C, Ferris LF, McCall L, Rommel N, van Wijk MP, Benninga MA, Moore D, Omari TI. Pressure-flow characteristics of normal and disordered esophageal motor patterns. J Pediatr. 2015 Mar;166(3):690-6.e1. doi: 10.1016/j.jpeds.2014.12.002. Epub 2015 Jan 13. PMID 25596103
- [Result] Omari T, Connor F, McCall L, Ferris L, Ellison S, Hanson B, Abu-Assi R, Khurana S, Moore D. A study of dysphagia symptoms and esophageal body function in children undergoing anti-reflux surgery. United European Gastroenterol J. 2018 Jul;6(6):819-829. doi: 10.1177/2050640618764936. Epub 2018 Mar 8. PMID 30023059
- [Result] Eckardt VF, Aignherr C, Bernhard G. Predictors of outcome in patients with achalasia treated by pneumatic dilation. Gastroenterology. 1992 Dec;103(6):1732-8. doi: 10.1016/0016-5085(92)91428-7. PMID 1451966
- [Result] Mellow MH, Pinkas H. Endoscopic therapy for esophageal carcinoma with Nd:YAG laser: prospective evaluation of efficacy, complications, and survival. Gastrointest Endosc. 1984 Dec;30(6):334-9. doi: 10.1016/s0016-5107(84)72448-5. PMID 6210226
- [Result] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151
- [Result] Omari TI, Szczesniak MM, Maclean J, Myers JC, Rommel N, Cock C, Cook IJ. Correlation of esophageal pressure-flow analysis findings with bolus transit patterns on videofluoroscopy. Dis Esophagus. 2016 Feb-Mar;29(2):166-73. doi: 10.1111/dote.12300. Epub 2014 Dec 17. PMID 25515292
- [Result] Lin Z, Imam H, Nicodeme F, Carlson DA, Lin CY, Yim B, Kahrilas PJ, Pandolfino JE. Flow time through esophagogastric junction derived during high-resolution impedance-manometry studies: a novel parameter for assessing esophageal bolus transit. Am J Physiol Gastrointest Liver Physiol. 2014 Jul 15;307(2):G158-63. doi: 10.1152/ajpgi.00119.2014. Epub 2014 May 22. PMID 24852565
- [Result] Omari TI, Papathanasopoulos A, Dejaeger E, Wauters L, Scarpellini E, Vos R, Slootmaekers S, Seghers V, Cornelissen L, Goeleven A, Tack J, Rommel N. Reproducibility and agreement of pharyngeal automated impedance manometry with videofluoroscopy. Clin Gastroenterol Hepatol. 2011 Oct;9(10):862-7. doi: 10.1016/j.cgh.2011.05.026. Epub 2011 Jun 6. PMID 21699810
- [Result] Omari TI, Dejaeger E, Van Beckevoort D, Goeleven A, De Cock P, Hoffman I, Smet MH, Davidson GP, Tack J, Rommel N. A novel method for the nonradiological assessment of ineffective swallowing. Am J Gastroenterol. 2011 Oct;106(10):1796-802. doi: 10.1038/ajg.2011.143. Epub 2011 May 10. PMID 21556039
- [Result] Myers JC, Nguyen NQ, Jamieson GG, Van't Hek JE, Ching K, Holloway RH, Dent J, Omari TI. Susceptibility to dysphagia after fundoplication revealed by novel automated impedance manometry analysis. Neurogastroenterol Motil. 2012 Sep;24(9):812-e393. doi: 10.1111/j.1365-2982.2012.01938.x. Epub 2012 May 23. PMID 22616652
- See also: Online tool for sharing manometry studies and performing P&F analysis — https://www.swallowgateway.com